CLINICAL TRIAL: NCT04295109
Title: Comparison of the Effects of Fentanyl, Oxycodone, Butorphanol on Gastrointestinal Function in Patients Undergoing Laparoscopic Hysterectomy: a Double-blind, a Randomized Controlled Trial
Brief Title: Comparison of the Effects of Fentanyl, Oxycodone, Butorphanol on Gastrointestinal Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shijiang Liu, Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2019-SR-476
Record Dates: First submitted 2020-01-05; First posted 2020-03-04 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cervix Neoplasms; Endometrial Cancer; Adenomyosis; Fibroid Uterus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Adenomyosis; Leiomyoma | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fentanyl group(group F) (Active Comparator): Fentanyl citrate injection, specification: 10mL: 0.5mg / piece (production unit: niching chang rendu Pharmaceutical Co., Ltd., valid period: 48 months) For group F patients,0.5mg fentanyl was mixed with saline to a total volume of 100mL; continuous infusion was set to 2mL/h, a bolus dose of 3mL, and a lockout interval of 15 minutes
  Interventions: Drug: the drug of intravenous patient-controlled analgesia
- Oxycodone group(group O) (Experimental): Oxycodone hydrochloride injection, specification: 1mL: 10mg / branch (production unit: HAMOL LIMITED, valid period: 60 months) For group O patients,30mg oxycodone was mixed with saline to a total volume of 100mL; continuous infusion was set to 2mL/h, a bolus dose of 3mL, and a lockout interval of 15 minutes
  Interventions: Drug: the drug of intravenous patient-controlled analgesia
- Butorphanol group(group B) (Experimental): Butorphanol tartrate injection, specification: 1 mL: 1 mg / branch (production unit: Jiangsu henryi Pharmaceutical Co., Ltd., valid period: 24 months); For group B patients,10mg butorphanol was mixed with saline to a total volume of 100mL; continuous infusion was set to 2mL/h, a bolus dose of 3mL, and a lockout interval of 15 minutes
  Interventions: Drug: the drug of intravenous patient-controlled analgesia

INTERVENTIONS:
Drug: the drug of intravenous patient-controlled analgesia — At present, opioids are most widely used in postoperative analgesia. This study aims to use different opioid receptor agonists---fentanyl, oxycodone and butorphanol for analgesia after laparoscopic hysterectomy.Compare the recovery of gastrointestinal function after operation.
  Other Names: intravenous patient-controlled analgesia (IV-PCA)

SUMMARY:
Postoperative ileus (POI) is a transient loss of coordinated peristalsis precipitated by surgery and exacerbated by opioid pain medication.So,how to provide patients with ideal analgesia without affecting the recovery of postoperative gastrointestinal function?This was a prospective randomized controlled study. A total of 105 patients who were scheduled for laparoscopic hysterectomy were randomly selected from The First Affiliated Hospital with Nanjing Medical University by random number table. These patients were randomly divided into three groups: fentanyl(F) group, oxycodone(O) group and butorphanol(B) group.

DETAILED DESCRIPTION:
Background: Patients often experience pain after gynecological laparoscopy. However, the use of opioid analgesia after surgery may increase the incidence of postoperative ileus (POI). Postoperative ileus (POI) is a common surgical emergency after a surgical procedure, leading to infection and intestinal adhesions, which can extend hospitalization and increase readmission rates, and consequently increasing healthcare costs. How to provide patients with ideal analgesia without affecting the recovery of postoperative gastrointestinal function? There is no guideline which has been troubling clinical anesthesiologists.

Aims: To observe the effects of fentanyl, oxycodone, Butorphanol on the recovery of gastrointestinal function after laparoscopic hysterectomy.

Methods: A total of 105 patients undergoing laparoscopic hysterectomy were randomly divided to three groups: fentanyl group(group F), butorphanol group(group B), or oxycodone group(group O). The primary outcome measures were postoperative time to first anal exhaust the total analgesic doses in PCIA,effective bolus times. Patients were also assessed for pain with a visual analogue scale (VAS), the cumulative PCIA dose, adverse effects (Nausea,vomiting, bradycardia, respiratory depression and pruritus), sedation level at 4, 12, 24, and 48 hours postoperatively, and satisfaction during the postoperative 48 hours and postoperative hospitalization days.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were scheduled for laparoscopic hysterectomy from W&C BRANCH HOSPITAL OF JIANGSU PROVINCE HOSPITAL
2. American Society of Anesthesiologists (ASA) physical status classification 1 to 2,
3. Women aged 40-65
4. Weight 50-80 kg

Exclusion Criteria:

1. History of opioids abuse and allergy and contraindication to opioid drugs
2. bronchial asthma; coronary heart disease; severe hypertension; diabetes mellitus;
3. hepatic, and renal dysfunction (glutamyl aminotransferase> 40U or aspartate aminotransferase> 35U; urea nitrogen> 8.2 μmol / L, creatinine> 133 μmol / L),
4. History of brain damage or psychiatric disease
5. Patients with coagulopathy (PT> 17 seconds or activated partial thromboplastin time (APTT)> 47 seconds);
6. pregnant or lactating women;
7. Those with long-term constipation;
8. History of digestive diseases;
9. history of gastrointestinal disease (peptic ulcer disease, Crohn's disease, or ulcerative colitis)
10. Participants in other drug trials in the past three months. （11）After randomization and allocation, patients were withdrawn if laparoscopy was converted to open surgery or if they required reinvestigation for postoperative bleeding.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
postoperative time to first anal exhaust | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 15 days
  Timing from the end of the operation
the cumulative dose administered in the patient-controlled mode | From date of operation until the date of first documented progression of anal exhaust , assessed up to 48 hours
  The cumulative dose administered in the patient-controlled mode during the initial 48 hours after the operation was measured
effective bolus times | From date of operation until the date of first documented progression of anal exhaust , assessed up to 48 hours
  The effective bolus times in the patient-controlled mode during the initial 48 hours after the operation was measured

SECONDARY OUTCOMES:
pain score | at 4 hours postoperatively
  by using numerical rating scale (NRS):The pain scale ranged from 0 (=no pain) to 10 (=worst pain imaginable)
pain score | at 12 hours postoperatively
  by using numerical rating scale (NRS):The pain scale ranged from 0 (=no pain) to 10 (=worst pain imaginable)
pain score | at 24 hours postoperatively
  by using numerical rating scale (NRS):The pain scale ranged from 0 (=no pain) to 10 (=worst pain imaginable)
pain score | at 48 hours postoperatively
  by using numerical rating scale (NRS):The pain scale ranged from 0 (=no pain) to 10 (=worst pain imaginable)
Sedation score | at 4 hours postoperatively
  by using Ramsay scale（1=anxious and agitated or restless, or both; 2=cooperative, oriented, and tranquil; 3=responds to command only; 4=asleep, but has a brisk response to light tactile stimulus or a simple verbal command; 5=asleep, but arousable only by strong physical stimulus; and 6=asleep, unarousable）
Sedation score | at 12 hours postoperatively
  by using Ramsay scale（1=anxious and agitated or restless, or both; 2=cooperative, oriented, and tranquil; 3=responds to command only; 4=asleep, but has a brisk response to light tactile stimulus or a simple verbal command; 5=asleep, but arousable only by strong physical stimulus; and 6=asleep, unarousable）
Sedation score | at 24 hours postoperatively
  by using Ramsay scale（1=anxious and agitated or restless, or both; 2=cooperative, oriented, and tranquil; 3=responds to command only; 4=asleep, but has a brisk response to light tactile stimulus or a simple verbal command; 5=asleep, but arousable only by strong physical stimulus; and 6=asleep, unarousable）
Sedation score | at 48 hours postoperatively
  by using Ramsay scale（1=anxious and agitated or restless, or both; 2=cooperative, oriented, and tranquil; 3=responds to command only; 4=asleep, but has a brisk response to light tactile stimulus or a simple verbal command; 5=asleep, but arousable only by strong physical stimulus; and 6=asleep, unarousable）
adverse effects | at 4 hours postoperatively
  Nausea 、vomiting 、bradycardia（HR <60 beats min-1）、respiratory depression(According to practice guidelines from the ASA, clinical signs of opioid-induced respiratory depression are respiratory rate <10 bpm, arterial O2 saturation <90%, or arterial CO2 tension >6.66 kPa) and pruritus
adverse effects | at 12 hours postoperatively
  Nausea 、vomiting 、bradycardia（HR <60 beats min-1）、respiratory depression(According to practice guidelines from the ASA, clinical signs of opioid-induced respiratory depression are respiratory rate <10 bpm, arterial O2 saturation <90%, or arterial carbon dioxide (CO2)tension >6.66 kPa) and pruritus
adverse effects | at 24 hours postoperatively
  Nausea 、vomiting 、bradycardia（HR <60 beats min-1）、respiratory depression (According to practice guidelines from the ASA, clinical signs of opioid-induced respiratory depression are respiratory rate <10 bpm, arterial O2 saturation <90%, or arterial CO2 tension >6.66 kPa)and pruritus
adverse effects | at 48 hours postoperatively
  Nausea 、vomiting 、bradycardia（HR <60 beats min-1）、respiratory depression (According to practice guidelines from the ASA, clinical signs of opioid-induced respiratory depression are respiratory rate <10 bpm, arterial O2 saturation <90%, or arterial CO2 tension >6.66 kPa)and pruritus
patients' degree of overall satisfaction with the postoperative analgesia | at 48 hours postoperatively
  Patients were asked to evaluate their degree of overall satisfaction with the postoperative analgesia on a 11-point scale (0= very unsatisfied, 1-3= unsatisfied, 4-6 = neutral, 7-9= satisfied, or 10 = very satisfied).
postoperative hospitalization days | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 15 days
  All patients were cured in accordance with clinical cure standard

CONTACTS AND LOCATIONS:
Overall Officials: Cunming Liu, doctorate, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Shijiang Liu, Master, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Chuanbao Han, Study Director — The First Affiliated Hospital with Nanjing Medical University; Minna Guo, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Guo M, Liu S, Gao J, Han C, Yang C, Liu C. The effects of fentanyl, oxycodone, and butorphanol on gastrointestinal function in patients undergoing laparoscopic hysterectomy: a prospective, double-blind, randomized controlled trial. BMC Anesthesiol. 2022 Feb 24;22(1):53. doi: 10.1186/s12871-022-01594-9. PMID 35209847